CLINICAL TRIAL: NCT00105131
Title: Genetic Characterization of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 050115; 05-N-0115
Record Dates: First submitted 2005-03-05; First posted 2005-03-07 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-11

CONDITIONS: Parkinson Disease; PD; Movement Disorder; Healthy Volunteer; HV
Keywords: Parkinson's Disease; Movement Disorders; Tremor; Alpha-Synuclein; Lewy Bodies; Parkinson Disease; PD; Movement Disorder; Healthy Volunteer; HV
MeSH Terms: conditions — Parkinson Disease; Movement Disorders; Tremor; Parkinson Disease 4, Autosomal Dominant Lewy Body

SUMMARY:
This study will explore the risks and causes of Parkinson's disease, a chronic progressive nervous system disorder. Patients typically have tremors, muscle weakness and a shuffling gait.

Patients with Parkinson's disease, their relatives and healthy volunteers may be eligible for this study. Candidates must be 18 years of age or older. Patients whose parkinsonism is due to a secondary cause, such as infection or injury, and healthy volunteers who have a first degree family member (parent, grandparent, child, sibling) with Parkinson's disease are excluded from enrollment.

Participants are asked about possible symptoms they may have and about their general health. They provide a blood sample to obtain DNA for genetic analysis to look for genetic differences that might be related to risks for Parkinson's disease. White blood cells may be treated in the laboratory to grow a cell line, which provides a source of substances in the blood without having to draw samples repeatedly.

DETAILED DESCRIPTION:
Parkinson's disease (PD) was noted to have a familial component as early as 1880. More recently, the discovery of several genetic factors influencing Parkinson's disease has emphasized the importance of heredity in PD.

Objective: The goal of this protocol will be to contribute to the genetic understanding of Parkinson's disease. Clinical data will be collected in order to document the features of Parkinson's disease in affected individuals (phenotyping). Genetic characterization will be undertaken for the discovery of specific genes which cause or contribute to the risk for Parkinson's disease (genotyping).

Design: The study design has two components. The first (aim 1) involves positional cloning for gene discovery in families with apparent Mendelian inheritance. The second (aim 2) will utilize an association study design, using genetic case-control methods for assessment of genetic risk factors. We will examine individuals affected by Parkinson's disease and their family members towards Specific Aim 1. Specific Aim 2 will involve evaluation of individuals with apparent sporadic Parkinson's disease, and also, healthy adult volunteers who will be recruited as control subjects.

Outcome Measures:

Primary Outcome Measures for Specific Aim 1 are:

1. The identification of new genes causal for Parkinson's disease.
2. The identification of new mutations in known genes.

Primary Outcome Measures for Specific Aim 2 are:

1. The discovery of gene variants which confer risk for Parkinson's disease.
2. The validation of already reported polymorphisms as risk factors for PD.

Secondary Outcome Measures (both Specific Aims 1 and 2): Genotype/phenotype correlations for specific genetic forms of Parkinson's disease. For example, we will assess if a particular age of onset, cardinal or secondary feature of PD or associated clinical course is associated with a given genotype.

Future Direction: Because 1) the larger sample base the greater the likelihood of the discovery of genes of minor effect and 2) discoveries of genetic risk factors require validation in additional sample series, it is likely that renewal of this protocol will be sought after five years.

Study Population: We aim to enroll a total of 2500 subjects over five years. These will include approximately 500 samples for the Mendelian studies (Specific Aim 1), and 2000 for association studies (Specific Aim 2). These estimates are based both on feasibility and on statistical power. Subjects will be evaluated at the NIH Clinical Center.

ELIGIBILITY:
INCLUSION CRITERIA:

Individuals with Parkinson's disease OR

Family members of an individual diagnosed with Parkinson's disease OR

Healthy adult controls obtained through the NIH Clinical Research Volunteers Program (CVRP) or other healthy control volunteers who come forward.

EXCLUSION CRITERIA:

Under the age of 18 years of age OR

Individuals with Parkinsonism secondary to a specific cause such as toxin exposure, birth injury, head injury, or brain infection such as encephalitis.

Healthy volunteers with a medical history or first degree family history of Parkinson's disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2500
Dates: Start 2005-03; Study Completion 2005-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Polymeropoulos MH, Lavedan C, Leroy E, Ide SE, Dehejia A, Dutra A, Pike B, Root H, Rubenstein J, Boyer R, Stenroos ES, Chandrasekharappa S, Athanassiadou A, Papapetropoulos T, Johnson WG, Lazzarini AM, Duvoisin RC, Di Iorio G, Golbe LI, Nussbaum RL. Mutation in the alpha-synuclein gene identified in families with Parkinson's disease. Science. 1997 Jun 27;276(5321):2045-7. doi: 10.1126/science.276.5321.2045. PMID 9197268
- [Background] Kitada T, Asakawa S, Hattori N, Matsumine H, Yamamura Y, Minoshima S, Yokochi M, Mizuno Y, Shimizu N. Mutations in the parkin gene cause autosomal recessive juvenile parkinsonism. Nature. 1998 Apr 9;392(6676):605-8. doi: 10.1038/33416. PMID 9560156
- [Background] Bonifati V, Rizzu P, van Baren MJ, Schaap O, Breedveld GJ, Krieger E, Dekker MC, Squitieri F, Ibanez P, Joosse M, van Dongen JW, Vanacore N, van Swieten JC, Brice A, Meco G, van Duijn CM, Oostra BA, Heutink P. Mutations in the DJ-1 gene associated with autosomal recessive early-onset parkinsonism. Science. 2003 Jan 10;299(5604):256-9. doi: 10.1126/science.1077209. Epub 2002 Nov 21. PMID 12446870